CLINICAL TRIAL: NCT05161143
Title: Efficacy and Safety of Donafenib Combined With TACE as Adjuvant Therapy of Patients With Hepatocellular Carcinoma at a High Risk of Recurrence After Radical Resection
Brief Title: Donafenib Combined With TACE as Adjuvant Therapy of Patients With Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SH3137
Record Dates: First submitted 2021-12-02; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; Adjuvant therapy; Donafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — donafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Donafenib plus TACE (Experimental): Donafenib: 4-8 weeks after radical surgery,patients will take donafenib, 200mg Bid,at least 6 months.
  TACE:4-8 weeks after radical surgery,Patients will receive TACE once.
  Interventions: Drug: Donafenib

INTERVENTIONS:
Drug: Donafenib — Donafenib: 4-8 weeks after radical surgery,patients will take donafenib, 200mg Bid,at least 6 months.
  TACE:4-8 weeks after radical surgery,patients will receive TACE once.
  Other Names: TACE

SUMMARY:
The investigators design a phase IIB clinical study to explore the efficacy and safety of Donafenib combined with TACE as adjuvant therapy of patients with hepatocellular carcinoma at a high risk of recurrence after radical resection.

DETAILED DESCRIPTION:
This trial is a single-arm, non-randomized and single-center clinical study of targeted therapy combined TACE in patients with hepatocellular carcinoma at a high risk of recurrence after radical resection.It is estimated that 30 patients who met the study criteria will be enrolled in Peking Union Medical College Hospital(PUMCH) and treated with Donafenib and TACE. The investigators will follow up and collect subjects' data monthly to evaluate the efficacy and safety of treatment, including overall survival and time to progression.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 ~ 75 years old (including boundary value), male and female;
2. Radical resection of liver cancer and intraoperative ablation of tumors ≤ 2cm were performed 4 ~ 8 weeks before enrollment;
3. Hepatocellular carcinoma diagnosed by pathology and meeting at least one of the following conditions:

   1. Single tumor with tumor size ≥ 5cm;
   2. Pathology showed microvascular invasion (MVI);
   3. Satellite foci were found in the specimens;
   4. Multiple lesions (≥ 3);
   5. AFP ≥ 400 ng / ml one week before operation
   6. Preoperative imaging and / or intraoperative or postoperative pathological reports found PVTT type I: tumor thrombus invaded the secondary and above branches of portal vein;
4. No anti-tumor treatment was received before operation;
5. Liver function grade child Pugh a;
6. Physical condition (PS) score of Eastern cancer cooperation group (ECoG) was 0-1;
7. Imaging examination ≥ 4 weeks after operation confirmed that there was no recurrence and metastasis;
8. The estimated survival time shall not be less than 3 months;
9. With sufficient organ function reserve, the laboratory test values within 14 days before treatment must meet the following standards:

   1. Blood routine examination: Hb≥100 g/L; ANC≥1.5 × 109 /L; PLT≥75 × 109 /L
   2. Biochemical examination: ALB ≥28g/L; ALT and AST < 5 × ULN; TBIL ≤2 × ULN; creatinine ≤ 1.5 × ULN or creatinine clearance (CCR) ≥ 50 ml / min
   3. The electrolyte is basically normal or normal after treatment;
   4. Urinary protein < 2 + or 24-hour urinary protein quantitative test ≤ 1.0 g / L (for patients with urinary protein ≥ 2 +, 24-hour urinary protein quantitative test should be carried out, and they can be selected only when it is ≤ 1.0 g / L);
   5. Coagulation function:

   international standard ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN activated partial coagulation time (APTT) ≤ 1.5 × ULN
10. Patients with HBsAg positive should continue antiviral treatment after operation and take first-line antiviral drugs such as entecavir or tenofovir or propofol tenofovir fumarate;
11. The patients were enrolled voluntarily, could provide written informed consent, and could understand and comply with the trial protocol to follow-up.

Exclusion Criteria:

1. The pathological diagnosis was fiberboard HCC, sarcomatoid HCC, hepatocellular carcinoma intrahepatic cholangiocarcinoma (HCC-ICC);
2. Positive margin or tumor rupture;
3. Reoperation of recurrent liver cancer;
4. Previous liver transplantation;
5. AFP did not return to normal at 4 weeks and did not return to normal at 6 weeks after operation;
6. Previously received systemic therapy for HCC, including targeted drug therapy such as Sorafenib, Lenvatinib and Regorafenib, or immunotherapy such as anti-PD-1, anti-PD-L1 and anti-CTLA-4, except antiviral therapy; If the patient has previously used traditional Chinese medicine with anti-tumor indications, it must be more than 4 weeks after the completion of treatment and before the medication in this study, and the adverse events caused by treatment have not recovered to ≤ CTCAE level 1;
7. Received other adjuvant therapy (except antiviral therapy), including adjuvant local therapy;
8. There were tumor thrombi in the main portal vein and primary branches, inferior vena cava, hepatic vein or bile duct, lymph node invasion or extrahepatic metastasis before operation;
9. 5 years of suffering from other malignancies, unless the patient has received the possibility of curative treatment and there is no evidence of the disease within 5 years, the time requirement (i.e. 5 years) does not apply to successful basal cell carcinoma, cutaneous squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ or other orthotopic cancer.
10. Previous history of severe mental illness;
11. Suffering from diseases affecting the absorption, distribution, metabolism or clearance of the study drug (such as severe vomiting, chronic diarrhea, intestinal obstruction, absorption disorder, etc.);
12. Taking drugs that may prolong QTc and / or induce tip twist transition ventricular tachycardia (TDP) or drugs that affect drug metabolism at the same time;
13. The patient has known or suspected allergy to tyrosine kinase inhibitor (TKI) drugs, or is allergic to the excipients of the study drugs;
14. There are uncontrollable hepatic encephalopathy, hepatorenal syndrome, ascites, pleural effusion or pericardial effusion;
15. Have active bleeding or abnormal coagulation function, have bleeding tendency or are receiving thrombolytic, anticoagulant or antiplatelet therapy;
16. Have a history of gastrointestinal hemorrhage or have a clear tendency of gastrointestinal bleeding in the past 4 weeks (e.g. local active ulcer lesions, fecal occult blood + + or more, gastroscopy should be performed if continuous fecal occult blood +, or other conditions that may cause gastrointestinal bleeding determined by the researcher (e.g. severe gastric fundus / esophageal varices);
17. Gastrointestinal perforation, abdominal fistula or abdominal abscess occurred in the past 6 months;
18. Thrombosis or thromboembolism events occurred in the past 6 months, such as stroke and / or transient ischemic attack, deep vein thrombosis, pulmonary embolism, etc;
19. Uncontrolled cardiovascular disease judged by the researcher. Including but not limited to the following situations:

    1. acute myocardial infarction in the past 6 months;
    2. Severe / unstable angina pectoris or coronary artery bypass grafting;
    3. Congestive heart failure (NYHA > 2);
    4. Arrhythmias with poor control or requiring pacemaker treatment;
    5. Hypertension (systolic blood pressure ≥ 140 mmHg and / or diastolic blood pressure ≥ 90 mmHg) ";
20. Active infection requiring treatment

    1. Active hepatitis B (HBsAg positive and abnormal liver function): if the HBV-DNA is ≥ 104 copies / ml within 14 days before treatment, the patient shall first undergo antiviral treatment, reduce it to < 104 copies / ml, and then enter the study, continue antiviral treatment and monitor liver function and serum HBV-DNA level;
    2. Active hepatitis C (HCV-RNA ≥ 103 copies / ml) with abnormal liver function [ALT or ast > 3 × ULN with TBIL > 2 × ULN or clinical jaundice]);
21. pregnant or lactating women, and female or male patients with fertility are unwilling or unable to take effective contraceptive measures;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
1 year RFS rate | 1 year
  1 year relapse-free survival rate

SECONDARY OUTCOMES:
RFS | 3 years
  Recurrence Free Survival
OS | 3 years
  Overall Survival
TTR | 3 years
  Time To Recurrence
2/3 year RFS rate | 2/3 years
  2/3 year Recurrence free survival rate
AE | 3 years
  Adverse events
AFP | 3 years
  Alpha fetal protein

CONTACTS AND LOCATIONS:
Overall Officials: Yilei Mao, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Global cancer statistics, 2002. CA Cancer J Clin. 2005 Mar-Apr;55(2):74-108. doi: 10.3322/canjclin.55.2.74. PMID 15761078
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Lu SD, Li L, Liang XM, Chen W, Chen FL, Fan LL, Ahir BK, Zhang WG, Zhong JH. Updates and advancements in the management of hepatocellular carcinoma patients after hepatectomy. Expert Rev Gastroenterol Hepatol. 2019 Nov;13(11):1077-1088. doi: 10.1080/17474124.2019.1684898. Epub 2019 Oct 30. PMID 31648568
- [Background] Akateh C, Black SM, Conteh L, Miller ED, Noonan A, Elliott E, Pawlik TM, Tsung A, Cloyd JM. Neoadjuvant and adjuvant treatment strategies for hepatocellular carcinoma. World J Gastroenterol. 2019 Jul 28;25(28):3704-3721. doi: 10.3748/wjg.v25.i28.3704. PMID 31391767
- [Background] Cucchetti A, Piscaglia F, Caturelli E, Benvegnu L, Vivarelli M, Ercolani G, Cescon M, Ravaioli M, Grazi GL, Bolondi L, Pinna AD. Comparison of recurrence of hepatocellular carcinoma after resection in patients with cirrhosis to its occurrence in a surveilled cirrhotic population. Ann Surg Oncol. 2009 Feb;16(2):413-22. doi: 10.1245/s10434-008-0232-4. Epub 2008 Nov 26. PMID 19034578
- [Background] European Association For The Study Of The Liver; European Organisation For Research And Treatment Of Cancer. EASL-EORTC clinical practice guidelines: management of hepatocellular carcinoma. J Hepatol. 2012 Apr;56(4):908-43. doi: 10.1016/j.jhep.2011.12.001. No abstract available. PMID 22424438
- [Background] Shen A, Liu M, Zheng D, Chen Q, Wu Z. Adjuvant transarterial chemoembolization after curative hepatectomy for hepatocellular carcinoma with microvascular invasion: A systematic review and meta-analysis. Clin Res Hepatol Gastroenterol. 2020 Apr;44(2):142-154. doi: 10.1016/j.clinre.2019.06.012. Epub 2019 Jul 11. PMID 31303533
- [Background] Ye JZ, Chen JZ, Li ZH, Bai T, Chen J, Zhu SL, Li LQ, Wu FX. Efficacy of postoperative adjuvant transcatheter arterial chemoembolization in hepatocellular carcinoma patients with microvascular invasion. World J Gastroenterol. 2017 Nov 7;23(41):7415-7424. doi: 10.3748/wjg.v23.i41.7415. PMID 29151695
- [Background] Wong JS, Wong GL, Tsoi KK, Wong VW, Cheung SY, Chong CN, Wong J, Lee KF, Lai PB, Chan HL. Meta-analysis: the efficacy of anti-viral therapy in prevention of recurrence after curative treatment of chronic hepatitis B-related hepatocellular carcinoma. Aliment Pharmacol Ther. 2011 May;33(10):1104-12. doi: 10.1111/j.1365-2036.2011.04634.x. Epub 2011 Mar 24. PMID 21488914
- [Background] Wu J, Yin Z, Cao L, Xu X, Yan T, Liu C, Li D. Adjuvant pegylated interferon therapy improves the survival outcomes in patients with hepatitis-related hepatocellular carcinoma after curative treatment: A meta-analysis. Medicine (Baltimore). 2018 Jul;97(28):e11295. doi: 10.1097/MD.0000000000011295. PMID 29995763
- [Background] Wang Z, Ren Z, Chen Y, Hu J, Yang G, Yu L, Yang X, Huang A, Zhang X, Zhou S, Sun H, Wang Y, Ge N, Xu X, Tang Z, Lau W, Fan J, Wang J, Zhou J. Adjuvant Transarterial Chemoembolization for HBV-Related Hepatocellular Carcinoma After Resection: A Randomized Controlled Study. Clin Cancer Res. 2018 May 1;24(9):2074-2081. doi: 10.1158/1078-0432.CCR-17-2899. Epub 2018 Feb 2. PMID 29420221
- [Background] Liu S, Guo L, Li H, Zhang B, Sun J, Zhou C, Zhou J, Fan J, Ye Q. Postoperative Adjuvant Trans-Arterial Chemoembolization for Patients with Hepatocellular Carcinoma and Portal Vein Tumor Thrombus. Ann Surg Oncol. 2018 Jul;25(7):2098-2104. doi: 10.1245/s10434-018-6438-1. Epub 2018 May 4. PMID 29728879
- [Background] Ono T, Yamanoi A, Nazmy El Assal O, Kohno H, Nagasue N. Adjuvant chemotherapy after resection of hepatocellular carcinoma causes deterioration of long-term prognosis in cirrhotic patients: metaanalysis of three randomized controlled trials. Cancer. 2001 Jun 15;91(12):2378-85. PMID 11413528
- [Background] Chen ZH, Zhang XP, Zhou TF, Wang K, Wang H, Chai ZT, Shi J, Guo WX, Cheng SQ. Adjuvant transarterial chemoembolization improves survival outcomes in hepatocellular carcinoma with microvascular invasion: A systematic review and meta-analysis. Eur J Surg Oncol. 2019 Nov;45(11):2188-2196. doi: 10.1016/j.ejso.2019.06.031. Epub 2019 Jun 25. PMID 31256949
- [Background] Wang L, Ke Q, Lin N, Zeng Y, Liu J. Does postoperative adjuvant transarterial chemoembolization benefit for all patients with hepatocellular carcinoma combined with microvascular invasion: a meta-analysis. Scand J Gastroenterol. 2019 May;54(5):528-537. doi: 10.1080/00365521.2019.1610794. Epub 2019 May 12. PMID 31081401
- [Background] Liao M, Zhu Z, Wang H, Huang J. Adjuvant transarterial chemoembolization for patients after curative resection of hepatocellular carcinoma: a meta-analysis. Scand J Gastroenterol. 2017 Jun-Jul;52(6-7):624-634. doi: 10.1080/00365521.2017.1292365. Epub 2017 Feb 22. PMID 28276833
- [Background] Wei W, Jian PE, Li SH, Guo ZX, Zhang YF, Ling YH, Lin XJ, Xu L, Shi M, Zheng L, Chen MS, Guo RP. Adjuvant transcatheter arterial chemoembolization after curative resection for hepatocellular carcinoma patients with solitary tumor and microvascular invasion: a randomized clinical trial of efficacy and safety. Cancer Commun (Lond). 2018 Oct 10;38(1):61. doi: 10.1186/s40880-018-0331-y. PMID 30305149
- [Background] Liu F, Guo X, Dong W, Zhang W, Wei S, Zhang S, Zhu X, Zhou W, Zhang J, Liu H. Postoperative adjuvant TACE-associated nomogram for predicting the prognosis of resectable Hepatocellular Carcinoma with portal vein Tumor Thrombus after Liver Resection. Int J Biol Sci. 2020 Oct 23;16(16):3210-3220. doi: 10.7150/ijbs.46896. eCollection 2020. PMID 33162826
- [Background] Huo YR, Chan MV, Chan C. Resection Plus Post-operative Adjuvant Transcatheter Arterial Chemoembolization (TACE) Compared with Resection Alone for Hepatocellular Carcinoma: A Systematic Review and Meta-analysis. Cardiovasc Intervent Radiol. 2020 Apr;43(4):572-586. doi: 10.1007/s00270-019-02392-6. Epub 2020 Jan 2. PMID 31897617
- [Background] Jiang H, Meng Q, Tan H, Pan S, Sun B, Xu R, Sun X. Antiangiogenic therapy enhances the efficacy of transcatheter arterial embolization for hepatocellular carcinomas. Int J Cancer. 2007 Jul 15;121(2):416-24. doi: 10.1002/ijc.22655. PMID 17330237
- [Background] Yao W, Xue M, Lu M, Wang Y, Zhao Y, Wu Y, Fan W, Li J. Diffuse Recurrence of Hepatocellular Carcinoma After Liver Resection: Transarterial Chemoembolization (TACE) Combined With Sorafenib Versus TACE Monotherapy. Front Oncol. 2020 Dec 17;10:574668. doi: 10.3389/fonc.2020.574668. eCollection 2020. PMID 33425729
- [Background] Chen JH, et al. 2020 ASCO. Poster 4580.
- [Background] Bruix J, Takayama T, Mazzaferro V, Chau GY, Yang J, Kudo M, Cai J, Poon RT, Han KH, Tak WY, Lee HC, Song T, Roayaie S, Bolondi L, Lee KS, Makuuchi M, Souza F, Berre MA, Meinhardt G, Llovet JM; STORM investigators. Adjuvant sorafenib for hepatocellular carcinoma after resection or ablation (STORM): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2015 Oct;16(13):1344-54. doi: 10.1016/S1470-2045(15)00198-9. Epub 2015 Sep 8. PMID 26361969